CLINICAL TRIAL: NCT01124630
Title: Pilot Study of CS-1008 in Combination With FOLFIRI (Irinotecan, Leucovorin, and 5-fluorouracil [5-FU]) in Subjects With Metastatic Colorectal Cancer (CRC) Who Have Failed First-line Treatment That Was Not Irinotecan-based.
Brief Title: Study of CS-1008 in Combination With FOLFIRI in Patients Who Have Failed Other Treatments
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS1008-A-U105
Record Dates: First submitted 2010-05-10; First posted 2010-05-17 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tigatuzumab; IFL protocol; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CS-1008 with FOLFIRI (Experimental): Experimental drug CS-1008 in combination with FOLFIRI
  Interventions: Drug: CS-1008; Drug: FOLFIRI

INTERVENTIONS:
Drug: CS-1008 — CS-1008 will be administered IV each week. The initial/loading dose (6 mg/kg) will be administered Day 1 of Cycle 1. Maintenance doses of 2 mg/kg will be administered weekly thereafter.
Drug: FOLFIRI — The FOLFIRI regimen will be administered IV at Weeks 1 and 3 of each 4 week cycle, and it will begin at Week 1 of Cycle 1. It will comprise irinotecan, 180 mg/m2 IV infusion over 30 to 120 minutes; leucovorin, 400 mg/m2 IV infusion to match the duration of the irinotecan infusion; and 5-FU, 400 mg/m2 (bolus) followed by 1200 mg/m2/day x 2 days (total 2400 mg/m2 over 46 to 48 hours continuous infusion).
  Other Names: irinotecan; leucovorin; 5-FU; Camptosar; Fluorouracil

SUMMARY:
Treatment with CS-1008 in combination with FOLFIRI (irinotecan, leucovorin, and 5-fluorouracil [5-FU]) in subjects with metastatic colorectal cancer (CRC) who have failed first-line treatment that was not irinotecan-based.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, metastatic CRC that has progressed after first-line standard therapy that was not irinotecan-based.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 2.
* Adequate organ and bone marrow function as evidenced by:

  * Hemoglobin >= 9 g/dL
  * White blood cell count (WBC) >= 3.0 x 109/L
  * Absolute neutrophil count (ANC) >= 1.5 x 109/L
  * Platelet count >= 100 x 109/L
  * Serum creatinine < the upper limit of normal (ULN)
  * AST and alkaline phosphatase =< 2.5 x ULN if without liver metastasis and =< 5.0 x ULN if liver metastasis
  * Total bilirubin =< ULN
* Male and female subjects of reproductive potential must be willing to consent to using effective contraception while on treatment and for 3 months after the end of treatment.
* Female subjects of childbearing potential must have a negative pregnancy test (serum or urine) result within 8 days before starting study treatment.
* Subjects must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an IRB-approved ICF before performance of any study-specific procedures or tests.
* At study centers located in the US, subjects must also sign a HIPAA authorization.
* KRAS Mutant

Exclusion Criteria:

* Anticipation of a need for a major surgical procedure or radiotherapy (RT) during the study.
* Treatment with chemotherapy, hormonal therapy, RT, minor surgery, or any investigational agent within 4 weeks before study enrollment. Treatment with nitrosoureas, mitomycin C, immunotherapy, biological therapy, or major surgery within 6 weeks before study enrollment.
* First-line therapy for CRC that was irinotecan-based.
* History of any of the following conditions within 6 months before study enrollment:

  * Myocardial infarction;
  * Severe/unstable angina pectoris;
  * Coronary/peripheral artery bypass graft;
  * New York Heart Association (NYHA) class III or IV congestive heart failure;
  * Cerebrovascular accident or transient ischemic attack;
  * Pulmonary embolism or other clinically significant thromboembolic event; or
  * Clinically significant pulmonary disease (eg, severe chronic obstructive pulmonary disease or asthma).
* Clinically active brain metastasis (ie, untreated, still requiring therapy with steroids or RT, or with progression within 4 weeks after completion of RT); an uncontrolled seizure disorder; spinal cord compression; or carcinomatous meningitis.
* History of malignancy other than CRC, unless there is the expectation that the malignancy has been cured, and tumor-specific treatment for the malignancy has not been administered within the previous 5 years.
* Clinically significant active infection that requires antibiotic therapy or Human Immunodeficiency Virus (HIV)-positive subjects receiving antiretroviral therapy.
* Previous treatment with CS-1008, other agonistic DRSantibodies, or with TRAIL agonists.
* If female, pregnant or breastfeeding.
* Known history of hypersensitivity reactions to any of the components of CS-1008, irinotecan, leucovorin, or 5-FU formulations.
* Serious intercurrent medical or psychiatric illnesses or any other conditions that in the opinion of the Investigator would impair the ability to give informed consent or unacceptably reduce protocol compliance or safety of the study treatment.
* Must not be known to be homozygous for the UGT1A1*28 allele, as this increases the risk for neutropenia following irinotecan treatment.
* Kras allele status must not be wild type.
* Dihydropyrimidine dehydrogenase (DPD) deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2010-05; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | up to 6 months
  To obtain a preliminary assessment of the antitumor activity of CS-1008 in combination with a FOLFIRI regimen based on the Objective Response Rate (ORR)
Progression Free Survival | up to 6 months
  To obtain a preliminary assessment of the antitumor activity of CS-1008 in combination with a FOLFIRI regimen based on the Progression Free Survival (PFS)

SECONDARY OUTCOMES:
Serum concentrations | weekly
  to determine serum concentrations at selected time intervals

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota